CLINICAL TRIAL: NCT01886222
Title: A Multi-center, Randomized, Controlled Trial to Evaluate the Efficacy and Safety of Long-term Mild Hypothermia in Adult Patients With Severe Traumatic Brain Injury
Brief Title: Randomized Controlled Trial of Long-term Mild Hypothermia for Severe Traumatic Brain Injury
Acronym: LTH-Ⅰ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); West China Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); The 101st Hospital of Chinese People's Liberation Army (Other); The 98 Hospital of People's Liberation Army (Unknown); Shenzhen Second People's Hospital (Other); The 94 Hospital of People's Liberation Army (Unknown); Nanfang Hospital, Southern Medical University (Other); The Affiliated Hospital of Medical College of Chinese People's Armed Police Forces (Unknown); Xiangya Hospital of Central South University (Other); Taizhou First People's Hospital (Other); Tang-Du Hospital (Other); Qilu Hospital of Shandong University (Other); Chongqing Emergency Medical Center (Other); Xuzhou Central Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Principal Investigator, Jiyao Jiang, Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RJNS001
Record Dates: First submitted 2013-06-17; First posted 2013-06-25 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Brain Injuries; Craniocerebral Trauma
Keywords: Traumatic brain injury
MeSH Terms: conditions — Brain Injuries; Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long-term mild hypothermia (Experimental): Focused intervention
  Interventions: Other: Long-term mild hypothermia
- Normothermia (Other): Standard management
  Interventions: Other: Normothermia

INTERVENTIONS:
Other: Long-term mild hypothermia — Hypothermia will be induced within 6 hours of injury and maintained at 34-35℃ for 5 days.Then the patients will be passively rewarmed to a temperature of 36 to 37˚C at a rate no greater than 0.5˚C/4 hours.
  Other Names: Mild hypothermia therapy
  Arms: Long-term mild hypothermia
Other: Normothermia — Patients assigned to the normothermia group will be kept at 36-37℃.
  Arms: Normothermia

SUMMARY:
This study is a prospective multi-centre randomized trial to compare the effect of long-term mild hypothermia versus routine normothermic intensive management in patients with severe traumatic brain injury.

The primary hypothesis is that the induction of mild hypothermia (maintained at 34-35℃) for 5 days will improve the outcome of patients at six months post injury compared with normothermia.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) remains a leading cause of death and disability in people with injuries and constitutes a major public health concern both in developed and developing countries. There are multiple clinical trials of hypothermia therapy for TBI conducted, however, with conflicting results. Subgroup analysis of most meta-analysis showed that therapeutic effect was significant when hypothermia was maintained more than 48 hours. We have previously reported a multicenter trial of mild hypothermia (33-35℃) for severe traumatic brain injury, in which 215 patients was randomized to long-term mild hypothermia group (n = 108) for 5 ±1.3 days mild hypothermia therapy and short-term mild hypothermia group ( n = 107) for 2±0.6 days mild hypothermia therapy. The results shown improved outcomes in patients with long-term mild hypothermia and similar frequency of complications. Therefore we concluded that long-term hypothermia, which maintains at 33-35℃ for 5 days, could be considered in the management of severe traumatic brain injury.

Hypothermia therapy was recommend as the level III evidence by the 2007 Brain Trauma Foundation's guideline and this treatment is currently used in our department and other large neurosurgical centers across China, with the aim to decrease the high intracranial pressure (ICP) and improve the functional outcome of TBI patients. When the decision was made, the injured patients would be placed on cooling blankets, tracheotomized and ventilated. The patients would receive continuous infusions of a paralytic drug (Tracrium 10-40 mg/hour) and chlorpromazine (5-10 mg/hour) administered using an infusion pump to prevent shivering. The dosage was given according to each patient's temperature, blood pressure, heart rate, and muscular tone. Once the patient's rectal temperature reached 33˚C, it was kept at approximately that temperature (33-35˚C) 5 to 7 days. Then the patients were passively rewarmed to a temperature of 37 to 38˚C at a rate no greater than 1˚C/hour, by gradual adjustment of the blanket thermostat.

The present multi-center, randomized controlled trials is designed to investigate the efficacy and safety of long-term (5 days) mild hypothermia versus normothermia on the outcome of patients following severe traumatic brain injury. The primary outcome is the neurological function assessed at 1, 6 months post injury with the Glasgow Outcome Score (GOS). Additionally, the following data will also be recorded and compared: the baseline data, Glasgow Coma Score,imaging examination (e.g. CT scan), need of surgery, intracranial pressure, laboratory tests (e.g. blood routine test, liver and kidney function, blood gas analysis, etc), the complications (e.g. pneumonia, significant bleeding) and so on.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years within 6 hours post injury;
* Closed head injury;
* Glasgow Coma Scale(GCS) score 4 to 8 after resuscitation;
* The intracranial pressure is more than 25 mmHg;
* Cerebral contusion on computed tomographic scan.

Exclusion Criteria:

* GCS of 3 with bilateral fixed and dilated pupils;
* A life-threatening injury to an organ other than the brain;
* No spontaneous breathing or cardiac arrest at the scene of the injury;
* No consent;
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Neurological function | 6 months post injury
  The neurological function will be evaluated at 6 months post injury by a specialized investigator who is unaware of the patients' allocation according to five-category Glasgow Outcome Scale as follows: 1, death; 2, vegetative state - unable to interact with the environment; 3, severe disability - unable to live independently but able to follow commands; 4, moderate disability - capable of living independently but unable to return to work or school; and 5, good recovery - able to return to work or school.

SECONDARY OUTCOMES:
Intracranial pressure (ICP) control | Admission, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 14, or until the monitor is removed
  The effect of long-term hypothermia on ICP control will be determined.
Glasgow Coma Score (GCS) | Admission, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 14, day 21, day 28 post injury
  The neurological function improvement during study intervention will be evaluated.
Length of ICU stay | 6 months post injury
  The numbers of days in the ICU.
Length of hospital stay | 6 months post injury
  The numbers of days in the hospital.
Frequency of complications | 6 months post injury
  Frequency of complications during the the study such as pneumonia, significant bleeding, liver and kidney function abnormality will be recorded and compared between groups.
Mortality rate | 6 months post injury
  The proportion of death will be determined at 6 months post injury.

CONTACTS AND LOCATIONS:
Overall Officials: Jiyao Jiang, MD, PhD, Principal Investigator — Department of Neurosurgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, China
Locations (1):
- Department of Neurosurgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Jiang JY, Xu W, Li WP, Gao GY, Bao YH, Liang YM, Luo QZ. Effect of long-term mild hypothermia or short-term mild hypothermia on outcome of patients with severe traumatic brain injury. J Cereb Blood Flow Metab. 2006 Jun;26(6):771-6. doi: 10.1038/sj.jcbfm.9600253. PMID 16306933
- [Background] Lei J, Gao G, Mao Q, Feng J, Wang L, You W, Jiang J; LTH-1 trial collaborators. Rationale, methodology, and implementation of a nationwide multicenter randomized controlled trial of long-term mild hypothermia for severe traumatic brain injury (the LTH-1 trial). Contemp Clin Trials. 2015 Jan;40:9-14. doi: 10.1016/j.cct.2014.11.008. Epub 2014 Nov 12. PMID 25460339
- [Derived] Hui J, Feng J, Tu Y, Zhang W, Zhong C, Liu M, Wang Y, Long L, Chen L, Liu J, Mou C, Qiu B, Huang X, Huang Q, Zhang N, Yang X, Yang C, Li L, Ma R, Wu X, Lei J, Jiang Y, Liu L, Gao G, Jiang J; LTH-1 Trial collaborators. Safety and efficacy of long-term mild hypothermia for severe traumatic brain injury with refractory intracranial hypertension (LTH-1): A multicenter randomized controlled trial. EClinicalMedicine. 2021 Jan 28;32:100732. doi: 10.1016/j.eclinm.2021.100732. eCollection 2021 Feb. PMID 33681741
- See also: Ren Ji Hospital is one of the top medical centers across China. — http://www.renji.com
- See also: Prof. Jiang holds the title of Chairman of International Neurotrauma Society. — http://www.neurotraumasociety.org/